CLINICAL TRIAL: NCT02838628
Title: A Phase 2a, Open-Label, Multicenter, Activity and Safety Study of KX2-391 Ointment 1% in Subjects With Actinic Keratosis on the Face or Scalp
Brief Title: Activity & Safety Study of KX2-391 Ointment in Participants With Actinic Keratosis on the Face or Scalp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KX01-AK-002; U1111-1173-5677 (Other: UTN)
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KX2-391 50 mg (Days 1 to 5) (Experimental): Participants were applied 50 milligrams (mg) of KX2-391 Ointment 1% topically on face or scalp in 25 centimeter square (cm^2) treatment area, once daily for 5 consecutive days.
  Interventions: Drug: 50 mg of KX2-391 Ointment 1%
- KX2-391 50 mg (Days 1 to 3) (Experimental): Participants were applied 50 mg of KX2-391 Ointment 1% topically on face or scalp in 25 cm^2 treatment area, once daily for 3 consecutive days.
  Interventions: Drug: 50 mg of KX2-391 Ointment 1%

INTERVENTIONS:
Drug: 50 mg of KX2-391 Ointment 1% — Dose: 50 mg; Route of administration: Topical
  Arms: KX2-391 50 mg (Days 1 to 5)
Drug: 50 mg of KX2-391 Ointment 1% — Dose: 50 mg; Route of administration: Topical
  Arms: KX2-391 50 mg (Days 1 to 3)

SUMMARY:
In this study, the activity, safety, and pharmacokinetics (PK) of KX2-391 Ointment was evaluated in adult participants with a clinical diagnosis of stable, clinically typical actinic keratosis (AK) on the face or scalp.

DETAILED DESCRIPTION:
This study was an open-label, multicenter, activity, safety, tolerability, and PK study of KX2-391 Ointment administered topically to the face or scalp of participants with AK.

The study consists of Screening, Treatment, and Follow-up Periods. Eligible participants were received 3 or 5 consecutive days of topical treatment, applied at the study site. Blood samples for PK analysis were collected. Activity (lesion counts) and safety evaluations were performed.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years old
2. Clinical diagnosis of stable, clinically typical actinic keratosis
3. A define treatment area on the face or scalp
4. Females must be postmenopausal, surgically sterile or otherwise incapable of pregnancy for at least 1 year; or must be using highly effective contraception for at least 90 days prior to treatment with KX2-391 Ointment
5. Males who have not had a vasectomy must agree to use barrier contraception
6. Participants who in the judgment of the Investigator, are in good general health
7. Willing to avoid excessive sun exposure
8. Able to comprehend and are willing to sign an informed consent form (ICF)

Exclusion Criteria:

1. Clinically atypical and/or rapidly changing AK lesions on the treatment area
2. Malignancy within 5 years prior to Screening except basal or squamous cell carcinoma not on the treatment area that were treated with curative intent and are without recurrence
3. Used any of retinoids at the most 90 days before Visit 1 glucocorticosteroids and methotrexate or other anti-metabolites within, at the most 28 days, before Visit 1
4. Used any topical therapies, treatments, or surgical or destructive modalities on the treatment area within, at the most 90 days, before Visit 1
5. Currently, or has experienced cutaneous malignancy, sunburn or body art on the treatment area within, at the most 180 days, before Visit 1
6. A history of sensitivity and/or allergy to any of the ingredients in the study medication
7. A skin disease or condition that, in the opinion of the Investigator, might interfere with the study conduct or evaluations, or which exposes the participant to an unacceptable risk by study participation
8. Other significant uncontrolled or unstable medical diseases or conditions that, in the opinion of the Investigator, would expose the participant to unacceptable risk by study participation
9. Females who are pregnant or nursing
10. Participated in an investigational drug trial during which an investigational study medication was administered within 14 days or 5 half-lives of the investigational product, whichever is longer, before dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Fang, MD, Study Chair — Kinex Pharmaceuticals Inc.
Locations (16):
- United States (16):
  - Center for Dermatology Clinical Research, Fremont, California
  - eStudy Site, La Mesa, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - International Dermatology Research, Miami, Florida
  - Compass Research, Orlando, Florida
  - Forward Clinical Trials, Inc., Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - Institute of Clinical Research - Tennessee, LLC, Murfreesboro, Tennessee
  - J&S Studies, Inc., College Station, Texas
  - The Center for Skin Research, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Dermatology Clinical Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kempers S, DuBois J, Forman S, Poon A, Cutler E, Wang H, Cutler D, Fang J, Kwan R. Tirbanibulin Ointment 1% as a Novel Treatment for Actinic Keratosis: Phase 1 and 2 Results. J Drugs Dermatol. 2020 Nov 1;19(11):1093-1100. doi: 10.36849/JDD.2020.5576. PMID 33196758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 sites in United States from 11 April 2016 to 22 December 2017.
Pre-assignment Details: A total of 168 participants (84 each cohort) were enrolled and treated in this study. This study consisted of 2 periods, first was Treatment and Follow-up period (up to Day 57) and second was Recurrence follow-up period (12 months post-Day 57).
Period: Treatment and Follow-up Period
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Started | 84 | 84
Completed | 84 | 84
Not Completed | 0 | 0
Period: Recurrence Follow-up Period
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Started (Participants who achieved 100% AK clearance at Day 57 visit entered the recurrence follow-up period.) | 36 | 27
Completed | 16 | 10
Not Completed | 20 | 17
Not completed — AK Recurrence | 18 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other un-specified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of study treatment.
Groups:
- KX2-391 50 mg (Days 1 to 5): Participants were applied 50 mg of KX2-391 Ointment 1% topically on face or scalp in 25 cm^2 treatment area, once daily for 5 consecutive days.
- Total: Total of all reporting groups
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3) | Total
Number analyzed (Participants) | 84 | 84 | 168
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (8.93) | 67.7 (8.32) | 68.3 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 76 | 72 | 148
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 81 | 75 | 156
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 84 | 83 | 167
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Number of AK Lesions [Mean (Standard Deviation); unit: Lesions] | 5.8 (1.41) | 5.4 (1.19) | 5.6 (1.32)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response of Actinic Keratosis
Description: Complete response rate was defined as the percentage of participants achieving 100% clearance in the treatment area on the face or scalp at Day 57.
Time Frame: Day 57
Population: Evaluable set included group of protocol-eligible participants who received 5 days (Cohort 1) or 3 days (Cohort 2) of study treatment and completed Day 1 and Day 57 AK lesion evaluations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
percentage of participants | 43 [32 to 54] | 32 [22 to 43]

2. Secondary Outcome: Percentage of Participants With Partial Response of Actinic Keratosis
Description: Partial response rate was defined as the percentage of participants achieving more than or equal to 75% clearance in the treatment area on the face or scalp at Day 57.
Time Frame: Day 57
Population: Per-protocol set included the group of protocol-eligible participants who received 5 days (Cohort 1) or 3 days (Cohort 2) of study treatment and completed at least one scheduled post treatment AK lesion evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
percentage of participants | 56 [45 to 67] | 52 [41 to 63]

3. Secondary Outcome: Overall Change From Baseline in Actinic Keratosis Lesion Counts at Day 8, 15, 29 and 57
Description: Overall changes from baseline in actinic keratosis lesion counts has been reported.
Time Frame: Baseline, Days 8, 15, 29 and 57
Population: as for outcome 2
Measure: Median (Full Range); unit: lesion count
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
lesion count
  Day 8 | 0.0 [-7 to 4] | -1.0 [-8 to 3]
  Day 15 | -2.5 [-8 to 5] | -2.0 [-8 to 2]
  Day 29 | -3.0 [-8 to 1] | -4.0 [-8 to 2]
  Day 57 | -4.0 [-8 to 1] | -4.0 [-8 to 0]

4. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an investigational Product (IP). An AE did not necessarily have a causal relationship with the medicinal product. An SAE was defined as any untoward medical occurrence that at any dose, resulted in death, was life-threatening (i.e, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). TEAEs were defined as either those AEs with an onset after dosing or those pre-existing conditions that worsened after dosing. TEAEs included both serious and non-serious TEAEs.
Time Frame: Baseline up to Day 57 (Treatment and follow-up period)
Population: Safety analysis set included group of participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
Participants | 34 | 18

5. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events During Recurrence Follow-up Period
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered an IP. An AE did not necessarily have a causal relationship with the medicinal product. An SAE was defined as any untoward medical occurrence that at any dose, resulted in death, was life-threatening (i.e, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). TEAEs were defined as either those AEs with an onset after dosing or those pre-existing conditions that worsened after dosing. TEAEs included both serious and non-serious TEAEs.
Time Frame: From Day 57 up to 12-months post-Day 57 (Recurrence follow-up period)
Population: Recurrence follow-up set included the group of participants who achieved complete clearance at Day 57.
Measure: Count of Participants; unit: Participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 36 | 27
Participants | 5 | 3

6. Secondary Outcome: Number of Participants With Maximal Post Baseline Local Skin Reactions (LSRs)
Description: Maximal post baseline LSR was defined as the highest grade of any LSR reported at any post baseline visits for a participant. Local skin reactions assessment included signs of erythema, flaking/scaling, crusting, swelling, vesiculation/pustulation, and erosion/ulceration on the treatment area. These signs were assessed using a 5-point grading scale ranging from 0 (not present) to 4 (worst), where (grade 0 = absent, grade 1 = slight, grade 2 = moderate, grade 3 = severe, grade 4 = very severe).
Time Frame: Day 57
Population: Safety analysis set included group of participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
Participants
  Erythema: LSR Grade 0 | 9 | 15
  Erythema: LSR Grade 1 | 22 | 34
  Erythema: LSR Grade 2 | 35 | 29
  Erythema: LSR Grade 3 | 17 | 6
  Erythema: LSR Grade 4 | 1 | 0
  Flaking/Scaling: LSR Grade 0 | 23 | 20
  Flaking/Scaling: LSR Grade 1 | 20 | 33
  Flaking/Scaling: LSR Grade 2 | 24 | 23
  Flaking/Scaling: LSR Grade 3 | 16 | 8
  Flaking/Scaling: LSR Grade 4 | 1 | 0
  Crusting: LSR Grade 0 | 49 | 53
  Crusting: LSR Grade 1 | 27 | 20
  Crusting: LSR Grade 2 | 8 | 10
  Crusting: LSR Grade 3 | 0 | 1
  Crusting: LSR Grade 4 | 0 | 0
  Swelling: LSR Grade 0 | 66 | 76
  Swelling: LSR Grade 1 | 16 | 8
  Swelling: LSR Grade 2 | 1 | 0
  Swelling: LSR Grade 3 | 1 | 0
  Swelling: LSR Grade 4 | 0 | 0
  Vesiculation/pustulation: LSR Grade 0 | 80 | 83
  Vesiculation/pustulation: LSR Grade 1 | 4 | 0
  Vesiculation/pustulation: LSR Grade 2 | 0 | 1
  Vesiculation/pustulation: LSR Grade 3 | 0 | 0
  Vesiculation/pustulation: LSR Grade 4 | 0 | 0
  Erosion/ulceration: LSR Grade 0 | 71 | 78
  Erosion/ulceration: LSR Grade 1 | 12 | 6
  Erosion/ulceration: LSR Grade 2 | 1 | 0
  Erosion/ulceration: LSR Grade 3 | 0 | 0
  Erosion/ulceration: LSR Grade 4 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory
Description: Laboratory parameters included hematology, blood chemistry and urinalysis. Clinical significance was determined by the investigator.
Time Frame: Baseline to Day 57
Population: Safety analysis set included group of participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs included measurement of pulse rate, systolic and diastolic blood pressure, respiratory rate, and body temperature. Clinical significance was determined by the investigator.
Time Frame: Baseline up to Day 57
Population: Safety analysis set included group of participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiograms (ECGs)
Description: ECG parameters included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals and corrected QT (QTc) intervals. Clinical significance was determined by the investigator.
Time Frame: Baseline up to Day 57
Population: Safety analysis set included group of participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
Participants | 4 | 1

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination (PE)
Description: A physical examination included weight and height measurements was performed. Clinical significance was determined by the investigator.
Time Frame: Baseline up to Day 57
Population: Safety analysis set included group of participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
Participants | 0 | 0

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of KX2-391 of KX2-391
Description: Cmax was defined as the maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1 and 4 hours post-dose on Days 1, 3 (Cohort 2) and 5 (Cohort 1)
Population: Pharmacokinetic (PK) Analysis Set included the group of participants who received study treatment and completed at least one scheduled post-treatment PK evaluation.
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
nanograms/milliliter (ng/mL) | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples. The maximum individual plasma concentration in both cohorts and all days of PK sampling did not exceed 2 ng/mL. | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples. The maximum individual plasma concentration in both cohorts and all days of PK sampling did not exceed 2 ng/mL.

12. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to the Last Sampling Time (AUCt) of KX2-391
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time (t) at which the concentration is at or above the LLOQ. AUC(0-t) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1 and 4 hours post-dose on Days 1, 3 (Cohort 2) and 5 (Cohort 1)
Population: PK Analysis Set included the group of participants who received study treatment and completed at least one scheduled post-treatment PK evaluation.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
nanogram*hour per milliliter (ng*h/mL) | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples. | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples.

13. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of KX2-391
Description: Cmin was defined as minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1 and 4 hours post-dose on Days 1, 3 (Cohort 2) and 5 (Cohort 1)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
ng/mL | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples. | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples.

14. Secondary Outcome: Accumulation Ratio (R)
Description: Ratio calculated from AUC and Cmax found on the last day of treatment and Day 1.
Time Frame: Pre-dose, 0.5, 1 and 4 hours post-dose on Days 1, 3 (Cohort 2) and 5 (Cohort 1)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
Number analyzed (Participants) | 84 | 84
ratio | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples. The maximum individual plasma concentration in both cohorts and all days of PK sampling did not exceed 2 ng/mL. | NA (NA) — Assessments of the PK parameters were planned but were not conducted due to the minimal absorption of KX2-391 in the plasma following 3 or 5 days of consecutive treatment of the 1% ointment. KX2-391 was below the lower limit of quantification (LLOQ) of 0.1 ng/mL for the majority of plasma samples. The maximum individual plasma concentration in both cohorts and all days of PK sampling did not exceed 2 ng/mL.

ADVERSE EVENTS:
Time Frame: Baseline up to Recurrence Follow-up (12 months post-day 57)
Description: Safety analysis set included group of participants who received at least one dose of study treatment.
Arm/Group | KX2-391 50 mg (Days 1 to 5) | KX2-391 50 mg (Days 1 to 3)
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84
Serious Adverse Events (participants affected / at risk) | 4/84 | 3/84
Other Adverse Events (participants affected / at risk) | 37/84 | 19/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KX2-391 50 mg (Days 1 to 5) (N=84) | KX2-391 50 mg (Days 1 to 3) (N=84)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1)
VIIth Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KX2-391 50 mg (Days 1 to 5) (N=84) | KX2-391 50 mg (Days 1 to 3) (N=84)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1) | 0 (0)
Defect Conduction Intraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Eye Discharge (Eye disorders) | 1 (1) | 0 (0)
Eye Pruritus (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Application Site Pain (General disorders) | 3 (3) | 2 (2)
Application Site Pruritus (General disorders) | 6 (7) | 1 (1)
Feeling Of Body Temperature Change (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dermatitis Contact (Immune system disorders) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Oral Herpes (Infections and infestations) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Electrocardiogram QT Prolonged (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscus Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Penile Ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Injury (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT02838628/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT02838628/SAP_001.pdf